CLINICAL TRIAL: NCT04054544
Title: A Gluten Challenge Study to Characterize Peripheral Blood and Intestinal Gluten-specific CD4+ T Cell Subsets in Patients With Celiac Disease
Brief Title: Gluten Challenge Study in Celiac Disease Participants (MK-0000-402)
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 0000-402; MK-0000-402 (Other: Merck)
Record Dates: First submitted 2019-08-05; First posted 2019-08-13 (Actual); Results first posted 2023-03-06 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2022-06

CONDITIONS: Celiac Disease
Keywords: Celiac disease
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Intervention Model Description: Experimental study to determine blood and duodenal T cell changes following administration of an 8 g gluten challenge daily for 13 days in participants with celiac disease
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gluten challenge (Experimental): Participants will receive a gluten 4 g powder twice daily (BID), for 13 consecutive days
  Interventions: Dietary Supplement: Gluten powder 4g

INTERVENTIONS:
Dietary Supplement: Gluten powder 4g — Gluten powder 4g oral BID

SUMMARY:
This is a gluten challenge study to characterize peripheral blood and intestinal gluten specific cluster of differentiation 4 glycoprotein (CD4+) thymus lymphocyte (T cell) subsets in participants with Celiac Disease

DETAILED DESCRIPTION:
This is a multi-site, open-label gluten challenge study to characterize peripheral blood and intestinal gluten specific CD4+ T cell subsets in participants with celiac disease (CeD). Participants will receive 8 grams (g) of gluten daily for 13 consecutive days. Blood samples will be taken at pre-dose, Day 6, and Day 14. Duodenal biopsy samples will also be collected on Day 14. Participants will also complete a symptom diary.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must have documented diagnosis with celiac disease (CeD) by duodenal/jejunal biopsy at least 6 months prior to entrance into the study.
2. Participant must be on a gluten-free diet (GFD) for at least the past 12 months.
3. Female participants must not be pregnant or breastfeeding. Women of childbearing potential (WOCBP) must use an acceptable contraceptive method or abstain from heterosexual intercourse.
4. Must be Human leukocyte antigen (HLA)-DQ2.5 positive, assessed at screening. If participants have already been genotyped, results from previous testing may be used in lieu of genotyping at screening.
5. Has anti-tissue transglutaminase (anti-tTG) <2x upper limit of normal (ULN) as measured by serology.
6. Be judged to be in good health based on medical history, physical examination (including a targeted neurological exam), versus (vs.) measurements and electrocardiogram (ECG) performed prior to treatment allocation.
7. Have a body mass index (BMI) 18-35 kg/m^2, inclusive.

Exclusion Criteria:

1. Has any chronic active gastrointestinal (GI) disease (e.g., clinically active CeD despite being on GFD for past 12 months, Crohn's disease, ulcerative colitis, lymphocytic colitis). Inactive, stable/well-treated lactose intolerance, Fermentable oligosaccharides, disaccharides, monosaccharides, and polyols (FODMAP) intolerance, gastroesophageal reflux disease (GERD), and irritable bowel syndrome (IBS) are allowed.
2. Has clinically active endocrine, gastrointestinal (other than CeD), cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, or major neurological (including stroke and chronic seizures) abnormalities or diseases. Participants with a remote history of uncomplicated medical events or stable medical diseases with no symptoms and stable treatment for the past >3 months may be enrolled in the study at the discretion of the investigator.
3. Is mentally or legally incapacitated, has significant emotional problems at the time of prestudy (screening) visit or expected during the conduct of the study or has a history of clinically significant psychiatric disorder within the last 5 years. Participants who have had situational depression may be enrolled in the study at the discretion of the investigator.
4. Participant has an estimated Glomerular Filtration Rate (eGFR) ≤80 mL/min/1.73 m^2 at the screening visit based on the Cockcroft-Gault (CG) equation
5. Has a history of significant multiple and/or severe allergies (e.g., food, drug, latex allergy), or has had an anaphylactic reaction or systemic allergic reaction to prescription or nonprescription drugs or food.
6. Subject has a history of severe acute symptomatic reactions to sporadic gluten ingestion.
7. Is positive for hepatitis B surface antigen, hepatitis C antibodies or human immunodeficiency virus (HIV).
8. Had major surgery, donated or lost 1 unit of blood (approximately 500 mL) within 4 weeks prior to the prestudy (screening) visit.
9. Is on Coumadin™ or other anticoagulants.
10. Is unable to refrain from or anticipates the use of systemic anti-inflammatory, immunosuppressive, or immunomodulatory medications, which may include ibuprofen > 2400 mg/day, naproxen >750 mg/day, prednisone >10 mg/day, or methylprednisolone > 8 mg/day, within 48 hours prior to the start of and throughout the entire gluten challenge.
11. Has participated in another investigational study within 4 weeks (or 5 half-lives, whichever is greater) prior to the prestudy (screening) visit. The window will be derived from the date of the last visit in the previous study.
12. Has a corrected QT (QTc) interval ≥470 msec (for males) or ≥480 msec (for females).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-08-28 (Actual); Primary Completion 2021-06-23 (Actual); Study Completion 2021-06-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (2):
- United States (2):
  - Massachusetts General Hospital ( Site 0001), Boston, Massachusetts
  - Beth Israel Deaconess Medical Center ( Site 0002), Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Groups:
- Gluten Challenge: Participants with celiac disease received 8 g gluten powder (4 g twice daily) orally for 13 consecutive days.
Period: Overall Study
Arm/Group | Gluten Challenge
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Gluten Challenge
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.9 (15.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of α1- and α2-gliadin-reactive CD4+ T Cells in Peripheral Blood Before Gluten Challenge
Description: Peripheral blood mononuclear cells (PBMC) collected prior to gluten challenge were stained with phycoerythrin (PE)-labeled human leukocyte antigen (HLA)-DQ2.5: gluten tetramers (DQ2.5-glia-α1 and DQ2.5-glia-α2) to identify antigen-specific cluster of differentiation (CD)4-positive thymus lymphocyte (T cells) reactive to gliadin (tetramer+ T cells) by flow cytometry. PBMC were also labeled with a 20-antibody panel for cell surface antigen staining to further define tetramer+ T cell subsets. Antigens included in the analysis were CD25, CD38, CD39, programmed cell death receptor 1 (PD-1), and integrin beta-7 (B7).
Time Frame: Baseline (Day 1, pre-dose)
Population: The analysis population includes participants who were compliant with study procedures and had available data.
Measure: Mean (Standard Deviation); unit: Percentage of T cells
Arm/Group | Gluten Challenge
Number analyzed (Participants) | 15
Percentage of T cells
  α1-gliadin tetramer+ | 0.00364 (0.00278)
  α1-gliadin tetramer+, CD25+ | 0.00016 (0.00029)
  α1-gliadin tetramer+, CD38+ | 0.00049 (0.00080)
  α1-gliadin tetramer+, CD39+ | 0.00005 (0.00021)
  α1-gliadin tetramer+, PD1+ | 0.00007 (0.00020)
  α1-gliadin tetramer+, Integrin B7+ | 0.00161 (0.00162)
  α2-gliadin tetramer+ | 0.01115 (0.00988)
  α2-gliadin tetramer+, CD25+ | 0.00058 (0.00092)
  α2-gliadin tetramer+, CD38+ | 0.00080 (0.00151)
  α2-gliadin tetramer+, CD39+ | 0.00006 (0.00024)
  α2-gliadin tetramer+, PD1+ | 0.00010 (0.00037)
  α2-gliadin tetramer+, Integrin B7+ | 0.00335 (0.00423)

2. Primary Outcome: Percentage of α1- and α2-gliadin-reactive CD4+ T Cells in Peripheral Blood After Gluten Challenge
Description: Peripheral blood mononuclear cells (PBMC) collected on Day 14 following gluten challenge were stained with phycoerythrin (PE)-labeled human leukocyte antigen (HLA)-DQ2.5: gluten tetramers (DQ2.5-glia-α1 and DQ2.5-glia-α2) to identify antigen-specific cluster of differentiation (CD)4-positive thymus lymphocyte (T cells) reactive to gliadin (tetramer+ T cells) by flow cytometry. PBMC were also labeled with a 20-antibody panel for cell surface antigen staining to further define tetramer+ T cell subsets. Antigens included in the analysis were CD25, CD38, CD39, programmed cell death receptor 1 (PD-1), and integrin beta-7 (B7).
Time Frame: Day 14
Population: The analysis population includes participants who were compliant with study procedures and had available data.
Measure: Mean (Standard Deviation); unit: Percentage of T cells
Arm/Group | Gluten Challenge
Number analyzed (Participants) | 15
Percentage of T cells
  α1-gliadin tetramer+ | 0.00707 (0.00510)
  α1-gliadin tetramer+, CD25+ | 0.00054 (0.00071)
  α1-gliadin tetramer+, CD38+ | 0.00276 (0.00161)
  α1-gliadin tetramer+, CD39+ | 0.00049 (0.00075)
  α1-gliadin tetramer+, PD1+ | 0.00091 (0.00113)
  α1-gliadin tetramer+, Integrin B7+ | 0.00361 (0.00198)
  α2-gliadin tetramer+ | 0.01315 (0.01199)
  α2-gliadin tetramer+, CD25+ | 0.00177 (0.00391)
  α2-gliadin tetramer+, CD38+ | 0.00495 (0.00698)
  α2-gliadin tetramer+, CD39+ | 0.00018 (0.00070)
  α2-gliadin tetramer+, PD1+ | 0.00186 (0.00378)
  α2-gliadin tetramer+, Integrin B7+ | 0.00609 (0.00470)

3. Primary Outcome: Percentage of α1-gliadin-reactive CD4+ T Cells in Duodenal Biopsies After Gluten Challenge
Description: Lymphocytes from duodenal biopsies collected on Day 14 following gluten challenge were stained with a phycoerythrin (PE)-labeled human leukocyte antigen (HLA)-DQ2.5: gluten tetramer (DQ2.5-glia-α1) to identify antigen-specific cluster of differentiation (CD)4-positive thymus lymphocyte (T cells) reactive to gliadin (tetramer+ T cells) by flow cytometry. Lymphocytes were also labeled with a 20-antibody panel for cell surface antigen staining to further define tetramer+ T cell subsets. Antigens included in the analysis were CD25, CD38, CD39, programmed cell death receptor 1 (PD-1), and integrin beta-7 (B7).
Time Frame: Day 14
Population: The analysis population includes participants who were compliant with study procedures and had available data.
Measure: Mean (Standard Deviation); unit: Percentage of T cells
Arm/Group | Gluten Challenge
Number analyzed (Participants) | 15
Percentage of T cells
  α1-gliadin tetramer+ | 0.29347 (0.26689)
  α1-gliadin tetramer+, CD25+ | 0.00263 (0.00401)
  α1-gliadin tetramer+, CD38+ | 0.19977 (0.19001)
  α1-gliadin tetramer+, CD39+ | 0.21248 (0.24696)
  α1-gliadin tetramer+, PD1+ | 0.26563 (0.26510)
  α1-gliadin tetramer+, Integrin B7+ | 0.24281 (0.24192)

ADVERSE EVENTS:
Time Frame: Up to 27 days
Description: All-cause mortality was analyzed in all randomized participants; Adverse events were analyzed in all randomized participants who received gluten challenge for at least one day.
Arm/Group | Gluten Challenge
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 16/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gluten Challenge (N=18)
Palpitations (Cardiac disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 10 (13)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 5 (6)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Epigastric discomfort (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Mucous stools (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 10 (11)
Rectal tenesmus (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (5)
Asthenia (General disorders) | 1 (1)
Fatigue (General disorders) | 9 (10)
Feeling abnormal (General disorders) | 4 (4)
Increased appetite (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Balance disorder (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 6 (6)
Insomnia (Psychiatric disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to unavailability of appropriate reagents, planned flow cytometry analyses of ω-gliadin reactivity and prevalence of CD95, tumor growth factor β1 receptor (TGFβ1R), and interleukin-27 receptor (IL-27R) antigens could not be performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor will generally support publication of multicenter studies only in their entirety and not as individual site data. In this case, a coordinating investigator will be designated by mutual agreement. If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-17): https://cdn.clinicaltrials.gov/large-docs/44/NCT04054544/Prot_SAP_000.pdf